CLINICAL TRIAL: NCT01582737
Title: Special Drug Use Investigation of Xarelto [SPAF]
Brief Title: Xarelto [SPAF] Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 15798; XAR-SPAF (Other: company internal)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Brain Ischemia
Keywords: Xarelto; SPAF
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with Xarelto for the purpose of prevention of ischemic stroke and systemic embolism
  Interventions: Drug: Rivaroxaban(Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban(Xarelto, BAY59-7939) — Patients treated with Xarelto under practical manner

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Xarelto for SPAF.

The objective of this study is to assess safety and effectiveness of Xarelto using in real clinical practice.

A total of 10,000 patients are to be enrolled and assessed in 2 years standard observational period. An annual follow-up survey will be conducted for 5 years at the longest after standard observational period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation (NVAF) for whom the decision to be treated with Xarelto was made
* Patients without experience of using Xarelto prior to the study

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-valvular arterial fibrillation necessary for the treatment for prevention of ischemic stroke and systemic embolism
Sampling Method: Non-Probability Sample
Enrollment: 11310 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs and serious AEs (especially for hemorrhagic events, and liver disfunction with increase of liver-function-relating enzymes including bilirubin) | Up to 2 years
Incidence of events of stroke | Up to 5 years
Incidence of events of non-central nervous system embolism | Up to 5 years

SECONDARY OUTCOMES:
Determination of patient's demography to affect the safety and efficacy of Xarelto using standard observational survey and follow-up survey | Baseline
Determination of patient's medical history to affect the safety and efficacy of Xarelto using standard observational survey and follow-up survey | Baseline
Determination of patient's background to affect the safety and efficacy of Xarelto using standard observational survey and follow-up survey | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Minematsu K, Ikeda T, Ogawa S, Kitazono T, Nakagawara J, Miyamoto S, Murakawa Y, Takeichi M, Kidani Y, Okayama Y, Sunaya T, Sato S, Yamanaka S. Real-World Outcomes of Rivaroxaban Treatment in Patients with Both Nonvalvular Atrial Fibrillation and a History of Ischemic Stroke/Transient Ischemic Attack. Cerebrovasc Dis. 2019;48(1-2):53-60. doi: 10.1159/000502883. Epub 2019 Oct 2. PMID 31578012
- [Derived] Ikeda T, Ogawa S, Kitazono T, Nakagawara J, Minematsu K, Miyamoto S, Murakawa Y, Iwashiro S, Kidani Y, Okayama Y, Sunaya T, Sato S, Yamanaka S. Outcomes associated with under-dosing of rivaroxaban for management of non-valvular atrial fibrillation in real-world Japanese clinical settings. J Thromb Thrombolysis. 2019 Nov;48(4):653-660. doi: 10.1007/s11239-019-01934-6. PMID 31432451
- [Derived] Nakagawara J, Ikeda T, Ogawa S, Kitazono T, Minematsu K, Miyamoto S, Murakawa Y, Takeichi M, Kidani Y, Okayama Y, Sunaya T, Sato S, Yamanaka S. Real-world outcomes of rivaroxaban treatment in patients with nonvalvular atrial fibrillation and worsening renal function. J Cardiol. 2019 Dec;74(6):501-506. doi: 10.1016/j.jjcc.2019.06.003. Epub 2019 Jul 29. PMID 31371191
- [Derived] Ikeda T, Ogawa S, Kitazono T, Nakagawara J, Minematsu K, Miyamoto S, Murakawa Y, Takeichi M, Ohashi Y, Okayama Y, Sunaya T, Yamanaka S. Real-world outcomes of the Xarelto Post-Authorization Safety & Effectiveness Study in Japanese Patients with Atrial Fibrillation (XAPASS). J Cardiol. 2019 Jul;74(1):60-66. doi: 10.1016/j.jjcc.2019.01.001. Epub 2019 Feb 8. PMID 30745002
- [Derived] Ogawa S, Minematsu K, Ikeda T, Kitazono T, Nakagawara J, Miyamoto S, Murakawa Y, Ohashi Y, Takeichi M, Okayama Y, Yamanaka S, Inuyama L. Design and baseline characteristics of the Xarelto Post-Authorization Safety & Effectiveness Study in Japanese Patients with Atrial Fibrillation (XAPASS). J Arrhythm. 2018 Feb 7;34(2):167-175. doi: 10.1002/joa3.12034. eCollection 2018 Apr. PMID 29657592